CLINICAL TRIAL: NCT04618276
Title: Effects of Photodynamic Therapy on the Human Inguinal Skin Microbiome to Improve Antiseptic Effect - Pilot 2
Brief Title: Effect of Photodynamic Therapy on Skin Microbiome. Single Center Study (PHOMIC-II)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020_PHOMIC-II
Record Dates: First submitted 2020-10-21; First posted 2020-11-05 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Postoperative Wound Infection Deep Incisional Surgical Site; Prosthesis and Implants; Surgical Site Infection; Prosthetic Joint Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Intervention group with PDT
  * Arm A will receive the photosensitizer 5-ALA
  * Arm B will receive Methylene blue as photosensitizer for the PDT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (5-ALA group) (Experimental): 1. Skin swab for culture in the groin for baseline
  2. PDT with 5% topical 5-ALA as the prodrug for the photosensitizer Pp IX
  3. Skin swab for culture
  4. Skin antisepsis
  5. Skin swab for culture
  Interventions: Other: Photodynamic Therapy
- Arm B (Methylene Blue group) (Experimental): 1. Skin swab for culture in the groin for baseline
  2. PDT with 0.01% methylene blue based photosensitizer (NF-031)
  3. Skin swab for culture
  4. Skin antisepsis
  5. Skin swab for culture
  Interventions: Other: Photodynamic Therapy
- Control group (No Intervention): 1. Skin swab for culture in the groin for baseline
  2. NO PDT
  3. Skin antisepsis
  4. Skin swab for culture

INTERVENTIONS:
Other: Photodynamic Therapy — PDT with two different photosensitizers
  Arms: Arm A (5-ALA group); Arm B (Methylene Blue group)

SUMMARY:
The overarching aim of this research project is to prevent orthopedic implant-associated infections. This study aims to investigate if PDT has an effect on bacterial skin colonization in order to improve skin antisepsis strategies for the prevention of surgical site infections.

DETAILED DESCRIPTION:
Background: Periprosthetic joint infections are a feared complication after orthopedic surgery in particular in our increasing elderly population. These infections are usually difficult to treat, because microorganisms persist in biofilms on the orthopedic implant surface. Therefore, it would be desirable to prevent these infections. It is hypothesized that bacteria from the skin surface or dermis - such as Staphylococcus aureus, coagulase-negative staphylococci, or Cutibacterium sp. - are transmitted into the periimplant tissue during surgery. In an ongoing interdisciplinary study with the Orthopedic University Hospital Balgrist (data in preparation for publication), the investigators see that common skin antisepsis preparation is not effective to eliminate skin bacteria before surgery because they persist in sebaceous or sweat glands. Photodynamic therapy (PDT) has recently gained attention in the treatment of acne, a disease of the pilosebaceous unit, in which also Cutibacterium acnes is implicated. The PDT works here on the one hand through a long-lasting destruction of the sebaceous glands, and on the other hand due to anti-inflammatory and antimicrobial effects.

In a previous pilot study, the investigators tested if skin antisepsis is improved with previous PDT with the photosensitizer-inducing prodrug 5% topical m5-aminolevulinic acid on inguinal skin in 10 participants. The induced photosensitizer was protoporphyrin IX (Pp IX, 635 nm) activated by red light. The investigators showed a complete sterilization of colonizing skin bacteria at the same day after this treatment However, orthopedic surgeons are hesitant to perform an arthroplasty surgery after such a treatment due to skin erythema for a few days.

The investigators are entirely convinced about this novel prevention concept but need to identify the photosensitizer with the ideal balance of antibactericidal effect versus skin irritation. Building upon the data they gathered, they will explore PDT with the Protoporphyrin IX inducing prodrug photosensitizer MAL and the photosensitizer Methylene blue with potentially less local side-effects (skin erythema).

Primary outcome:

Effect of photodynamic treatment with the photosensitizers Pp IX (5-ALA) and Methylene blue in combination with surgical antisepsis on bacterial skin colonization on the day of application and on day 1, 3, and 5 after PDT.

Secondary outcome:

Effect of PDT on the skin microbiome using molecular techniques.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants ≥ 18 years who

  * volunteer for the pilot study in which a routine photodynamic treatment in the Department of Dermatology will be applied and effect of skin colonization will be analyzed, and
  * an informed consent is signed by the participant (after information about the project).

Exclusion Criteria:

* Pregnant and lacting women
* Participants with inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.,
* Participants taking antibiotics in the 14 days prior to PDT or until follow-up at 21 days
* Participants who received oral retinoid therapy within the last 6 months
* Participants who received anti-inflammatory agents as NSAR within the 14 days prior and after the PDT
* Participants taking any photosensitizing drugs within 4 weeks prior to PDT
* Participants who had a history of photosensitivity disorder
* Fitzpatrick's skin phototype V-VI

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Each study participant was a control participant as well (procedure on the contralateral leg without intervention)
Units Other Than Participants: PDT: right side, no PDT left side
Groups:
- Arm A (MAL Group): 1. Skin swab for culture in the groin for baseline
  2. PDT with 5% topical methyl aminolevulinate (MAL) as the prodrug for the photosensitizer Pp IX
  3. Skin swab for culture
  4. Skin antisepsis
  5. Skin swab for culture
  Photodynamic Therapy: PDT with two different photosensitizers
- Arm B (Methylene Blue Group): 1. Skin swab for culture in the groin for baseline
  2. PDT with 0.01% methylene blue based photosensitizer (NF-031)
  3. Skin swab for culture
  4. Skin antisepsis
  5. Skin swab for culture
  Photodynamic Therapy: PDT with two different photosensitizers
Period: Overall Study
Arm/Group | Arm A (MAL Group) | Arm B (Methylene Blue Group)
Started (Each of the 10 participant was his own control. We performed PDT on the right leg and on the left leg no PDT (control)) | 10; 20 PDT: right side, no PDT left side | 10; 20 PDT: right side, no PDT left side
Completed (Each participant was his own control (no PDT on the contralateral leg)) | 10; 20 PDT: right side, no PDT left side | 10; 20 PDT: right side, no PDT left side
Not Completed | 0; 0 PDT: right side, no PDT left side | 0; 0 PDT: right side, no PDT left side

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (MAL Group) | Arm B (Methylene Blue Group) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 27.5 [19 to 36] | 32 [19 to 59] | 30 [19 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With no Growth of Bacteria on the Skin
Description: Quantitative evaluation of bacterial density and species from skin swabs taken before PDT, immeadiately after PDT, and after after skin antisepsis using culture technique
Time Frame: Day 0 after PDT
Population: Number of patients with no growth of bacteria on the skin
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (MAL Group) | Arm B (Methylene Blue Group)
Number analyzed (Participants) | 10 | 10
Participants
  PDT group right side | 3 | 7
  Control side without PDT | 6 | 7

2. Primary Outcome: Number of Patients With no Growth of Bacteria on the Skin on After 1 Day
Description: Quantitative evaluatuation of bacterial density and species from skin swabs taken 1 day after PDT before and after skin antisepsis
Time Frame: Day 1 after PDT
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (5-ALA Group): 1. Skin swab for culture in the groin for baseline
  2. PDT with 5% topical 5-ALA as the prodrug for the photosensitizer Pp IX
  3. Skin swab for culture
  4. Skin antisepsis
  5. Skin swab for culture
  Photodynamic Therapy: PDT with two different photosensitizers
Arm/Group | Arm A (5-ALA Group) | Arm B (Methylene Blue Group)
Number analyzed (Participants) | 10 | 10
Participants | 2 | 7

3. Primary Outcome: Number of Patients With no Growth of Bacteria on the Skin After 3 Days
Description: Quantitative evaluatuation of bacterial density and species from skin swabs taken 3 days after PDT before and after skin antisepsis
Time Frame: Day 3 after PDT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (5-ALA Group) | Arm B (Methylene Blue Group)
Number analyzed (Participants) | 10 | 10
Participants | 3 | 6

4. Primary Outcome: Number of Patients With no Growth of Bacteria on the Skin on Day 5 Number of Patients With no Growth of Bacteria on the Skin on Day 5
Description: Quantitative evaluatuation of bacterial density and species from skin ...
Time Frame: Day 5
Population: Day 5 was for most of the patients on the weekend which was not feasible to take swabs. Therefore we skipped day 5
Arm/Group | Arm A (5-ALA Group) | Arm B (Methylene Blue Group)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Arm A (MAL Group) | Arm B (Methylene Blue Group) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/20
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT04618276/Prot_SAP_000.pdf